CLINICAL TRIAL: NCT02239757
Title: Left vs Right Radial Approach in the Setting of Primary Percutaneous Coronary Intervention for ST-elevation Myocardial Infarction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Buxing Chen, Director of department of cardiology, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LERRASMI; Lerrasmi (Registry Identifier: Lerrasmi)
Record Dates: First submitted 2014-09-11; First posted 2014-09-15 (Estimated); Last update posted 2015-08-03 (Estimated); Status verified 2014-09

CONDITIONS: Transradial Approach, Primary PCI, ST-segment Elevation Myocardial Infarction
Keywords: Transradial Approach, Primary PCI, ST-segment elevation myocardial infarction
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Right radial approach (Experimental): Primary PCI performed through right radial approach.
  Interventions: Procedure: Left radial approach
- Left radial approach (Experimental): Primary PCI performed through left radial approach.
  Interventions: Procedure: Right radial approach

INTERVENTIONS:
Procedure: Left radial approach — Primary PCI performed through left radial approach.
  Arms: Right radial approach
Procedure: Right radial approach — Primary PCI performed through right radial approach.
  Arms: Left radial approach

SUMMARY:
Outcomes of patients with acute ST-elevation myocardial infarction (STEMI) are directly related to reperfusion time. Effect of transradial approach (left vs right) on reperfusion time has not been fully studied for SETMI patients undergoing primary percutaneous coronary intervention (PCI). The aim of this study was to randomly investigate the efficacy and safety of left radial approach for primary PCI in STEMI patients compared with right radial approach.

DETAILED DESCRIPTION:
The investigators will enroll consecutively for 3 years all STEMI patients undergoing primary PCI.

Patients will be included within 12 hours of symptom onset for primary PCI. Patients will be excluded if they are in cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

All consecutive patients with ST-segment elevation myocardial infarction within 12 hours of symptom onset for primary PCI.

Exclusion Criteria:

Patients are excluded if they were in cardiogenic shock.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2013-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Needle to balloon time | 1 day

SECONDARY OUTCOMES:
Radiation dose | 7 days
  Radiation dose include cumulative air kerma (CAK) and CAK dose area product (CAK DAP)
Fluoroscopy time | 7 days
Contrast volume | 7 days

OTHER OUTCOMES:
Vascular complications | 7 days
  Vascular complications include pseudoaneurysm, arteriovenous fistula, lose of radial artery pulse, puncture site bleeding and forearm hematoma.

CONTACTS AND LOCATIONS:
Overall Officials: Buxing Chen, MD, Ph.D, Principal Investigator — Beijing Tiantan Hospital
Locations (1):
- Beijing Tiantan Hospital, Capital Medical University, Beijing, China

REFERENCES:
- [Background] Hu H, Fu Q, Chen W, Wang D, Hua X, Chen B. A prospective randomized comparison of left and right radial approach for percutaneous coronary angiography in Asian populations. Clin Interv Aging. 2014 Jun 20;9:963-8. doi: 10.2147/CIA.S64235. eCollection 2014. PMID 25018624